CLINICAL TRIAL: NCT02707588
Title: A Phase II Randomized Study to Determine the Tolerance and Efficacy of Pembrolizumab or Cetuximab Combined With Radiation Therapy in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Tolerance and Efficacy of Pembrolizumab or Cetuximab Combined With RT in Patients With Locally Advanced HNSCC
Acronym: PembroRad
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2015-01
Record Dates: First submitted 2016-02-29; First posted 2016-03-14 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2022-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Determine the tolerance and efficacy of Pembrolizumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Antibodies; Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pembrolizumab and radiotherapy (Experimental): 200 mg IV infusion every 3 weeks, i.e. on day 1, 22, 43 during the course of radiotherapy
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy
- Cetuximab and radiotherapy (Active Comparator): Loading dose of 400 mg/m² IV on Day-8, followed by weekly dose of 250 mg/m² IV during the whole course of radiotherapy.
  Interventions: Drug: Cetuximab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — 200mg IV infusion every 3 weeks, i.e. on day 1, 22, 43 during the course of radiotherapy.
  Radiotherapy will be delivered daily for 5 days per week to a total dose of 69.96 Gy in 2.12 Gy daily fractions over 6.5 weeks (33 fractions).
  Other Names: antibody
  Arms: Pembrolizumab and radiotherapy
Drug: Cetuximab — Loading dose of 400 mg/m² IV on Day-8, followed by weekly dose of 250 mg/m² IV during the whole course of radiotherapy.
  Radiotherapy will be delivered daily for 5 days per week to a total dose of 69.96 Gy in 2.12 Gy daily fractions over 6.5 weeks (33 fractions).
  Other Names: antibody
  Arms: Cetuximab and radiotherapy
Radiation: Radiotherapy — Radiotherapy will be delivered daily for 5 days per week to a total dose of 69.96 Gy in 2.12 Gy daily fractions over 6.5 weeks (33 fractions).
  Other Names: Conventional Radiotherapy

SUMMARY:
The general aim of the study is to evaluate the anti-tumour activity and the tolerance profile of Pembrolizumab + RT in comparison to cetuximab + RT in patients with locally advanced HNSCC and to explore potential correlations between treatment outcome and the immune landscape.

DETAILED DESCRIPTION:
A majority of HNSCC are locally advanced and commonly treated with concomitant chemo-radiotherapy (CT-RT). However, a large proportion of patients with locally advanced stage are not suitable for receiving cisplatinum-based chemotherapy (CT) concomitant with radiotherapy (RT) either due to age, general and/or medical condition(s).

An alternative standard treatment has been established, combining RT and cetuximab.

However, both CT-RT and cetuximab-RT which are considered as standard approaches in locally advanced non operated HNSCC are associated with poor outcome in patients with the most advanced T stage (T4) and/or N stage (>=N2) and/or HPV negative tumours. A new and promising approach could target immune response.

Pembrolizumab is a high-affinity monoclonal anti-PD1 antibody which showed antitumor activity in melanoma and NSCLC. In the KEYNOTE-012 (multi-center, nonrandomized Phase Ib HNSCC), Pembrolizumab was well tolerated and safe with no serious drug related AEs reported. About 51% (26/51) of patients had decreased tumor burden which was seen both in HPV (-) and HPV(+) HNSCC.

This observation led to the hypothesis generated in the current study that Pembrolizumab is potentially a very active drug in HNSCC and that the combination of Pembrolizumab with radiotherapy will be well tolerated, given the very good toxicity profile of the drug and will improve the outcome of patients with locally advanced HNSCC non suitable for CT-RT, as compared to the treatment of reference combining cetuximab and RT.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥18 ≤ 80 years.
3. Performance Status ECOG 0-1
4. Histologically confirmed diagnosis of previously untreated locally advanced HNSCC (Stage III, IVa and IVb according to the American Joint Committee on Cancer Staging System) of one or more of the following sites: oral cavity, oropharynx, hypopharynx and larynx
5. Availability of pre-treatment tumour tissue (for biomarker analysis, PD -L1, TILs and immune-monitoring)
6. p16 expression from tumor sample (immunohistochemistry)
7. Recording of the smoking history
8. No viral infection (HIV, Hepatitis B/C)
9. No autoimmune disease
10. No immunodeficiency or immunosuppressive therapy
11. No active CNS disease
12. No interstitial lung disease
13. No active infection
14. Women of child-bearing potential: negative serum pregnancy test at screening and use of appropriate contraception methods from study entry
15. Patients not proposed cisplatin-based chemotherapy because of age, general condition, if medically unfit or patient refusal.
16. Adequate organ laboratory values
17. Health insurance coverage

Exclusion Criteria:

1. Nasopharyngeal, paranasal sinuses, nasal cavity tumours or thyroid cancers;
2. Squamous cell cancer involving cervical neck nodes with unknown primary site;
3. Metastatic disease;
4. Any prior or current treatment for invasive head and neck cancer. This will include but is not limited to: prior tyrosine kinase inhibitors, any monoclonal antibody, prior neoadjuvant therapy, prior surgical resection, or use of any investigational agent;
5. Weight loss of >10% during the last 3 weeks prior the screening visit;
6. Concurrent treatment with any other systemic anti-cancer therapy that is not specified in the protocol;
7. Concomitant treatment with any drug on the prohibited medication list such as live vaccines (for details, see the protocol);
8. History of another malignancy within the last 3 years (exception of in situ carcinoma and skin carcinomas);
9. If female, pregnant or lactating;
10. Significant disease which, in the judgment of the investigator, as a result of the medical interview, physical examinations, or screening investigations would make the patient inappropriate for entry into the trial.
11. Known hypersensitivity reaction to study medication;
12. Any social, personal, medical and/or psychologic factor(s) that could interfere with the observance of the patient to the protocol and/or the follow-up and/or the signature of the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Locoregional Control | 15 months from the end of radiation therapy
  To compare between the 2 arms the rate of patients achieving Locoregional Control (LRC) at 15 months from the end of radiation therapy

SECONDARY OUTCOMES:
Progression free survival | At 24 months after treatment initiation
  Minimum time from randomization to progression/relapse at any site (local, regional or distant) as defined by RECIST 1.1 criteria or to death from any cause. Patients who don't have any of these events are censored at the date of last follow-up.
Locoregional progression and distant metastasis | At 24 months after treatment initiation
  To estimate the respective contribution of locoregional progression, distant progression and death as first event in the progression-free survival, the cumulative incidences of these three types of events were calculated within a competing risk framework.
Overall survival | At 24 months after treatment initiation
  Time to death from any cause measured from randomization.
Acute adverse events | At 24 months after treatment initiation
  According to NCI-CTCAE version 4, the maximal grade of each toxicity observed during immune-radiotherapy will be used. All grades of toxicity will be tabulated by type of toxicity and by treatment arm.
Delayed toxicity According to RTOG late toxicity scale | At 24 months after treatment initiation
  According to RTOG late toxicity scale
Duration of the feeding tube dependence | At 24 months after treatment initiation
  It will be presented by treatment arm and analysed by Student t-test.
Compliance to Pembrolizumab and Cetuximab | At 24 months after treatment initiation
  Insufficient compliance to cetuximab or Pembrolizumab is defined as a patient receiving less than 75% of the planned dose, even if the dose reduction is due to toxicity
Health related quality of life (QL) | At 24 months after treatment initiation
  Assessment by EORTC QLQ-C30 and H&N35 questionnaires
Impact of p16 / HPV tumor status on the efficacy of the 2 regimens in patients with oropharyngeal initial tumor | At 24 months after treatment initiation
  Assessment by CISH DNA method

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pr BOURHIS, MD, Principal Investigator — CHU Vaudois, Rue du Bugnon 46, CH-1011 Lausanne, Suisse
Locations (1):
- Centre Guillaume le conquérant, Le Havre, France

IPD SHARING:
Plan to Share IPD: Yes